CLINICAL TRIAL: NCT03702738
Title: A Prospective Randomized Controlled Trial of Adjunctive N-acetylcysteine (NAC) in Adult Patients With Pulmonary Tuberculosis: a Sub-study of TB Sequel
Brief Title: Adjunctive NAC in Adult Patients With Pulmonary Tuberculosis
Acronym: NAC-TB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Aurum Institute NPC (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUR1-1-219
Record Dates: First submitted 2018-10-04; First posted 2018-10-11 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Host-directed therapy; N-acetylcysteine; Glutathione
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC (Experimental): Patients will be randomized to receive standard TB treatment with N-acetylcysteine 1200 mg BID x 4 months, followed by 2 months of standard TB treatment alone
  Interventions: Drug: N-acetyl cysteine
- No NAC (No Intervention): Patients will be randomized to receive 6 months standard TB treatment alone

INTERVENTIONS:
Drug: N-acetyl cysteine — NAC is listed by WHO as an essential medicine for its use in paracetamol (acetaminophen) poisoning, in which it protects against fatal liver injury. It also reduces the viscosity of sputum, thereby serving as an expectorant.
  Other Names: NAC
  Arms: NAC

SUMMARY:
To determine if adjunctive N-acetylcysteine 1200 mg twice a day (BID) accelerates sputum culture conversion and normalization of cellular glutathione in tuberculosis (TB), and to assess its potential effects on lung and immune function

DETAILED DESCRIPTION:
This is a randomized controlled, 2-arm, parallel group substudy of the TB-SEQUEL cohort study. It will enrol drug sensitive TB patients with moderately advanced or far advanced pulmonary disease by chest X-ray. Patients providing informed consent will undergo screening evaluations to establish eligibility. Patients meeting all the inclusion and none of the exclusion criteria will be randomized to receive standard TB treatment (2HRZE/4HR) plus NAC 1200 mg BID for months 1-4, or standard treatment alone. During the treatment period patients will undergo safety, efficacy, and biomarker assessments at specified time points. After a final evaluation at 6 months, patients will continue follow-up as a part of the main TB-SEQUEL cohort study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years, male or female
2. Willing and able to provide signed written consent or witnessed oral consent in the case of illiteracy, prior to undertaking any trial related procedures.
3. Body weight (in light clothing without shoes) between 40 and 90 kg.
4. First episode of pulmonary tuberculosis
5. Positive sputum AFB smear with subsequent culture confirmation OR positive Xpert TB/RIF with Ct ≤27.1 [3].
6. RIF susceptibility diagnosed by Xpert TB/RIF OR Hain test
7. Chest radiograph meeting criteria for moderate or far advanced pulmonary tuberculosis [4]
8. If sexually active, willing to use an effective contraceptive method for the duration of tuberculosis treatment
9. HIV-1 seronegative, or if HIV-1 seropositive, CD4 T cell count >220/ul

Exclusion Criteria:

1. Any condition for which participation in the trial, as judged by the investigator, could compromise the well being of the subject or prevent, limit or confound protocol specified assessments
2. Current or imminent (within 24 hr) treatment for malaria.
3. Pregnancy
4. Is critically ill, and in the judgment of the investigator has a diagnosis likely to result in death during the trial or the follow up period.
5. TB meningitis or other forms of severe tuberculosis with high risk of a poor outcome as judged by the investigator.
6. History of allergy or hypersensitivity to any of the trial therapies or related substances, including known allergy or suspected hypersensitivity to rifampin.
7. Having participated in other clinical trials with investigational agents within 8 weeks prior to trial start or currently enrolled in an investigational trial.
8. Prior TB treatment in the preceding 6 months.
9. Angina pectoris requiring treatment with nitroglycerin or other nitrates
10. Cardiac arrhythmia requiring medication, or any clinically significant ECG abnormality, in the opinion of the investigator
11. Random blood glucose >140 mg/dL, or history of unstable Diabetes Mellitus which required hospitalization for hyper- or hypo-glycaemia within the past year prior to start of screening.
12. Use of systemic corticosteroids within the past 28 days.
13. Patients requiring treatment with medications not compatible with rifampin, such as HIV-1 protease inhibitors
14. Subjects with any of the following abnormal laboratory values:

    1. creatinine >2 mg/dL
    2. haemoglobin <8 g/dL
    3. platelets <100x109 cells/L
    4. serum potassium <3.5
    5. aspartate aminotransferase (AST) ≥2.0 x ULN
    6. alkaline phosphatase (AP) >5.0 x ULN
    7. total bilirubin >1.5 mg/dL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Median time to stable sputum culture conversion using liquid medium | 6 months

SECONDARY OUTCOMES:
Change from baseline in mean concentration of reduced glutathione (GSH) in blood cells, expressed as the AUC during days 1-28 | 1-28 days
GSH concentrations and the ratio of GSH to GSSG (oxidized glutathione) measured at discrete time points during treatment | 6 months
Whole blood bactericidal activity (WBA) prior and at intervals post dosing | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wallis, Principal Investigator — Chief Scientific Officer
Locations (1):
- NIMR-Mbeya Medical Research Centre, Mbeya, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wallis RS, Sabi I, Lalashowi J, Bakuli A, Mapamba D, Olomi W, Siyame E, Ngaraguza B, Chimbe O, Charalambous S, Rachow A, Ivanova O, Zurba L, Myombe B, Kunambi R, Hoelscher M, Ntinginya N, Churchyard G. Adjunctive N-Acetylcysteine and Lung Function in Pulmonary Tuberculosis. NEJM Evid. 2024 Sep;3(9):EVIDoa2300332. doi: 10.1056/EVIDoa2300332. Epub 2024 Aug 27. PMID 39189858